CLINICAL TRIAL: NCT05517499
Title: Efficacy of Dexamethasone in Treatment of Meconium Aspiration Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB/2021/771/SIMS
Record Dates: First submitted 2022-05-20; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Efficacy, Self
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Dexamethasone Group), (Experimental): Group A (Case Group) was given dexamethasone i.e., 0.2 mg per kg per day every 12 hours for 7 days intravenously. All treatment strategies were same in both groups but steroid was given to group A
  Interventions: Drug: Dexamethasone
- Group B (Control Group) (No Intervention): Group B (Control group), received routine treatment.No dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Randomized clinical trial
  Other Names: no dexamethasone
  Arms: Group A (Dexamethasone Group),

SUMMARY:
Objective: To determine efficacy of dexamethasone in treatment of meconium aspiration syndrome.

Study design: Randomized control trial. Place and duration: Services hospital, Neonatal unit, Lahore. During time span of 1st January to 30th June 2021.

Material and methods Total 100 neonates were randomly divided in two groups. Group A (n=50) was treated with dexamethasone (Cases) and Group B (n=50) served as control. Dexamethasone was given in dose of 0.2mg/kg, 12 hourly for 7 days after confirmation of diagnosis. Infants present in clinical trial were evaluated by ventilation duration (invasive and non-invasive), oxygen therapy and hospital stay.

DETAILED DESCRIPTION:
Data was analyzed in statistical analysis SPSS version 23. Means and Standard deviation were calculated for duration of non-invasive and invasive ventilation, hospital stay and oxygen therapy. Independent sample T test was applied and value < 0.05 was taken as significant. Whereas frequency and percentages were taken for gender, gestation, mode of delivery and outcome of MAS and Chi-square test was applied, and p value < 0.05 was taken as significant.

ELIGIBILITY:
Inclusion Criteria:

1. Term and Post-Term babies who met the operational definition of MAS (inborn)
2. Presenting within 24 hours of life

Exclusion Criteria:

1. Preterm babies or babies with congenital malformations
2. Preterm babies or babies with dysmorphism
3. Preterm babies or babies with hypoxic-ischemic encephalopathy

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
The number of days required for ventilation in participants | 7 days
  The purpose of study was to measure number of days required for ventilation in participants
The number of days required for oxygen therapy in participants | 7 days
  The purpose of study was to measure number of days required for oxygen therapy in participants
The number of days required for hospitalization in participants | 7 days
  The purpose of study was to measure number of days required for hospitalization in participants

CONTACTS AND LOCATIONS:
Overall Officials: Uzair Qureshi, FCPS, Study Chair — Services Institute of Medical Sciences, Pakistan
Locations (1):
- Services Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No